CLINICAL TRIAL: NCT07283471
Title: Enriching Relational Environments by Using Purposeful Interactions and Building Developmental Relationships With Children in Out of Home Care
Brief Title: Facilitating Developmental Interactions With Children in Out-of-Home Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 141953; R01HD109329 (NIH)
Record Dates: First submitted 2025-12-11; First posted 2025-12-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Psychological Trauma
Keywords: trauma; children; out-of-home care
MeSH Terms: conditions — Psychological Trauma; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The intervention is a workshop that includes two sessions for staff and supervisors together and two additional sessions just for supervisors. The goal of the workshop series is to help staff and supervisors who care for children in residential settings learn how to provide more developmentally enriching interactions for the children in their care, who frequently suffer from the effects of maltreatment and/or neglect or other adverse childhood experiences. For these children, the accumulation of consistent interactions with adults who are attuned to the child's needs and feelings, listen to and respect those needs and feelings, and help the children learn to cope with those needs and feelings provide pathways to more normative developmental trajectories.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Developmental Interaction Workshop Series (Other): The two-part Developmental Interactions Workshop series is designed for adults who work with children in out-of-home care settings and the people who supervise these adults. Part 1 and Part 2 of this series include two sessions each: one session for direct caregivers and their supervisors, and one additional session for supervisors only. Part 2 of the workshop series should take place 3-4 weeks after Part 1.
  The focus of these workshops is helping caregivers to take advantage of the everyday and ordinary moments in daily life to create developmental interactions with children that help the child feel connected to others, capable, and autonomous. Supervisor only sessions will focus on the ways in which they can support and assist their staff to intentionally create these moments with children.
  Interventions: Behavioral: The Developmental Interaction Workshop Series (DIWS)

INTERVENTIONS:
Behavioral: The Developmental Interaction Workshop Series (DIWS) — Many children living in out-of-home care have experienced ongoing trauma, toxic stress, and adversity. These experiences have had a significant impact on children's ability to regulate their feelings and behaviors, enjoy healthy relationships, and grow along typical developmental pathways. To help these children to begin to heal from their past experiences and resume a more typical developmental trajectory, they need repetitive developmentally enriching interactions with adult caregivers. This requires caregivers with the willingness and ability to engage in frequent daily interpersonal exchanges with children that meet their emerging developmental needs and strengthen their internal resources to engage, grow, and heal. The DIWS is designed to help caregivers take advantaqe of the everyday and ordinary moments in daily life to create developmental interactions with children that help the child feel connected to others, capable, and autonomous.

SUMMARY:
The first goal of this single arm clinical trial is to develop the Developmental Interactions Workshop Series (DIWS). The second goal is to learn about the DIWS's acceptability, feasibility, and usefulness by implementing it in agencies who provide residential care for children.

The main questions it answers are

* Does participating in the DIWS help caregivers to become more capable, motivated, and purposeful about using developmental interactions in their caregiving role?
* Do caregivers and children see more developmental interactions during their routine daily activities after the caregivers complete the DIWS?

Caregiving staff will

* Attend the DIWS
* Complete surveys 2-4 before and 4-6 weeks after the DIWS
* Complete telephone interviews before and after the DIWS (a subset of caregiving staff)

Children in care will complete brief surveys 2-4 weeks before and 4-8 weeks after their caregiving staff attend the DIWS.

DETAILED DESCRIPTION:
Most U.S. children living in residential care (RC) have debilitating impairments regulating emotions and behavior and the success of treatment efforts for these children depends principally on caregivers' capacity to provide developmentally enriching, therapeutic care. While living in RC, the adults who care for these children during the critical hours outside of formal therapy play central roles in their treatment. Yet, RC caregivers receive little education about how to meet the unique relational needs of the children they serve and lack a clear understanding of their own therapeutic role in each child's rehabilitation. In addition, the most commonly-used training programs for caregivers in RC, as well as other out-of-home care settings, cover an eclectic range of topics without a specific focus on relational skills, and few have empirical support. Ultimately, in order for RC services to optimize children's rehabilitation and mitigate the long-term sequelae of developmental trauma, it is imperative to provide opportunities for caregivers to develop skills for eliciting developmentally enriching interactions (DIs) during their ordinary care routines. Toward that goal, the investigators propose two specific aims. Aim #1: Produce a video-based Developmental Interaction Workshop Series (DIWS) that enables caregivers to repeatedly observe and practice specific forms of DI and to create opportunities to increase their frequency during daily care routines. The DIWS will include two 4-hour sessions for caregivers and supervisors together, as well as one 2-hour and one 3-hour session for supervisors. A beta version will be implemented in one Residential Care (RC) agency, revised as needed, and then fully implemented in at least two RC agencies. Aim #2: Evaluate the DIWS using mixed methods (staff and child surveys, staff interviews, and ethnography) in 2-4 RC agencies to document preliminary evidence of its impact, acceptability, and feasibility. The investigators expect the DIWS to lead (1) caregivers to become more capable, motivated, and purposeful about eliciting DIs in their caregiving role, and (2) caregivers and children to perceive a greater prevalence of DIs during routine daily activities. Individual, organizational, and implementation-related factors related to uptake will also be identified. The DIWS will provide a developmentally-informed framework for understanding and enhancing the child-adult relationships in residential and other out-of-home care settings. Mixed-method evaluation results will provide the foundation for future RCTs of the program's efficacy, inform program improvements, and facilitate its wider dissemination.

ELIGIBILITY:
Inclusion Criteria

* Residential care staff in agencies participating in the Developmental Interactions Workshop Series
* Children 8 years of age or older living in agencies participating in the Developmental Interactions Workshop Series

Exclusion Criteria

• Children 7 years of age or younger living in agencies participating in the Developmental Interactions Workshop Series

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Frequency of Caregiving Practices over the past week from prior to attending the Developmental Interaction Workshop Series to 4 weeks after the final workshop | From completion of the staff survey 2 weeks prior to the initial workshop to 4 weeks after the final workshop. The two parts of the workshop are delivered 3-4 weeks apart.
  This self-report measure of staff practices is adapted for the residential child care setting from the Involvement subscale of the Alabama Parenting Questionnaire (Shelton, Frick, & Wootton, 1996, Journal of Clinical Child Psychology, 253:317-329). The 7-point response scale for each of the 13 items ranges from 0=not at all to 6=Very Often, yielding overall scores ranging from 0=not at all to 78=very often on all items with higher numbers indicating more positive practices.

SECONDARY OUTCOMES:
Change in commitment to the goal of increasing developmental interactions currently, from before attending the Developmental Interaction Workshop Series to 4 weeks after the final workshop | From completion of the staff survey 2 weeks prior to the initial workshop to 4 weeks after the final workshop. The two parts of the workshop are delivered 3-4 weeks apart.
  This self-report measure Goal Commitment is adapted for the current program goal from the Goal Commitment Scale (Klein, H. J., Wesson, M. J., Hollenbeck, J. R., Wright, P. M., & DeShon, R. P. (2001). Organizational Behavior and Human Decision Processes, 85(1), 32-55. The 5 point response scale on which respondents rate their agreement with the four items ranges from 0 =Not at all to 4=Completely yielding scores ranging from 0 to 16 with higher numbers indicating higher commitment.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Sellers, PhD, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No
The DIWS will be completed at 2-3 agencies that provide residential treatment for children. Given the magnitude of the commitment to implementing the Developmental Interaction Workshop Series at an agency, it is not possible to fully guarantee masking the agencies who participate. Thus, the potential to identify individuals in participant data is increased, particularly if information (staff versus supervisor, age and gender of the child) crucial to proper use of the data is included.

REFERENCES:
- [Background] Klein HJ, Wesson MJ, Hollenbeck JR, Wright PM, DeShon RP. The Assessment of Goal Commitment: A Measurement Model Meta-Analysis. Organ Behav Hum Decis Process. 2001 May;85(1):32-55. doi: 10.1006/obhd.2000.2931. PMID 11341816
- [Background] Shelton, K. K., Frick, P. J., & Wootton, J. (1996). Assessment of parenting practices in families of elementary school-age children. Journal of clinical child psychology, 25(3), 317-329.